CLINICAL TRIAL: NCT01672333
Title: Phase 2 Study of Response Rate and Side Effects of Preoperative Chemotherapy With Docetaxel, Oxaliplatin and Capcitabine (TOX) in Patients With Locally Advanced Operable Gastric Adenocarcinoma
Brief Title: Response Rate and Side Effects of Preoperative Chemotherapy (TOX Regimen) in Patients With Locally Advanced Operable Gastric Adenocarcinoma
Acronym: TOX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Milad Hospital (Other)
Responsible Party: Principal Investigator, Dr Seyed-Hossein Yahyazadeh-Jabari, Director of Clinical Research Center, Milad Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOX protocol
Record Dates: First submitted 2012-08-14; First posted 2012-08-24 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pathological Response (Experimental)
  Interventions: Drug: TOX

INTERVENTIONS:
Drug: TOX — oxaliplatin 100mg/m2 IV over 2 hours at 1st day docetaxel 50 mg/m2 IV over 1 hour at 1st day capecitabine 625 mg/m2 PO for 14 days

SUMMARY:
Early stage diagnosis of gastric cancer has ensued different approaches in its resection strategies. In order to increase the proportion of cases that undergo radical resection and reduce the recurrence rate, different pre-operative treatments are introduced. Here, the investigators investigate an active preoperative chemotherapeutic regimen to in patients with locally advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Tissue diagnosis of gastric or gastroesophageaql junction Adenocarcinoma
* T3, T4 any N with non metastatic condition
* Age 18 - 70 years
* Performance status 0,1 according to ECOG criteria
* Adequate bone marrow , liver and renal function
* Hemoglobin ≥ 11 g/dl
* Platelets ≥ 100000 / mm3
* Absolute Neutrophil Count ≥ 1500/mm3
* Normal Bilirubin
* Normal Transaminases
* Normal creatinin
* Absence of active co-morbid illness (uncontrolled infection, uncontrolled DM, cardiopulmonary disease)

Exclusion Criteria:

* Any metastatic disease, T1, T2, N0

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-06; Primary Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Pathologic Response rate | Participants are assessed after 4 chemotherapy courses 3 weeks apart, an expected period of 12 weeks from starting the study treatment protocol.
  A single expert pathologist evaluates the pathologic outcome of the chemotherapy regimen after the completion of courses. Participants are divided into 3 groups including complete pathologic response, partial pathologic response and pathologic stable disease.

SECONDARY OUTCOMES:
clinical Response rate | Participants are assessed after 2 courses of Chemotherapy 3 weeks apart, an expected period of 6 weeks from starting the study treatment protocol.
  A single expert clinician evaluates the clinical outcome of the chemotherapy regimen after 2 primary courses 3 weeks apart. Evaluation is done with regards to the "TNM" scoring of gastric cancer (T for the size and expansion of the tumor, N for lymph node involvement, M for distant metastasis). Participants are divided into 4 groups including clinically progressive disease, complete clinical response, partial clinical response and clinically stable disease.

CONTACTS AND LOCATIONS:
Overall Officials: Bahram Salmanian, M.D., Principal Investigator — Milad Hospital
Locations (1):
- Fayyazbakhsh hospital, Tehran, Tehran Province, Iran